CLINICAL TRIAL: NCT02712437
Title: Prospective Study Evaluating the Use of PROSPECT, a Cognitive Behavioral Therapy-based Internet Module, to Reduce Insomnia in Patients With Early Stage Breast Cancer
Brief Title: Prospective Study Evaluating the Use of PROSPECT to Reduce Insomnia in Patients With Early Stage Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of low accrual.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2015.168
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer; Insomnia
Keywords: Insomnia; Quality of Life; Cognitive behavioral therapy
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PROSPECT (Experimental): Participants who have received treatment for early stage breast cancer and who experience chronic insomnia as assessed by difficulty sleeping for >30 days with an insomnia severity index score of >14. Participants will complete baseline symptom questionnaires and actigraphy, then complete an internet-based cognitive behavioral therapy program (PROSPECT) for 6 weeks. Participants will then repeat questionnaires and actigraphy at 6 weeks and questionnaires at 12 weeks.
  Interventions: Behavioral: PROSPECT

INTERVENTIONS:
Behavioral: PROSPECT — PROSPECT is an internet-based exercise and behavioral symptom management program developed for patients who experience long-term side effects from cancer treatment. The cancer-specific symptom management intervention is intended as a self-management adjunct to improve cancer- and treatment-related symptoms, including insomnia, through non-pharmacologic approaches.

SUMMARY:
Women with early stage breast cancer may experience difficulty falling asleep or staying asleep. If this occurs for more than 4 weeks, these participants may have chronic insomnia. Chronic insomnia can lead to difficulty coping with stress, changes in mood, increased use of medications for sleep and an overall decrease in quality of life.

The investigators have developed an internet-based website that is designed to help people manage symptoms typically experienced by breast cancer survivors, including insomnia, fatigue, pain and overall poor quality of life. The investigators want to learn whether this type of treatment can reduce chronic insomnia and improve the way subjects feel using both questionnaires and a special form of a wrist watch. This information may help the investigators better manage sleep difficulties in subjects who experience these symptoms after diagnosis of their breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of insomnia as identified through the screening Insomnia Severity Index score >14
2. Insomnia present for > 30 days per patient report
3. Female gender
4. Histologically proven stage 0-III invasive carcinoma of the breast

   a. Patient's must have completed primary surgical resection at least 2 weeks prior to enrollment, radiation at least 2 weeks prior to enrollment and/or cytotoxic chemotherapy at least 6 weeks prior to enrollment in the study
5. ECOG performance status 0-2
6. Ability to operate the accelerometer (Actiwatch Spectrum Pro)
7. The patient is aware of the nature of her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent document

Exclusion Criteria:

1. Subjects who do not have access to the internet to use the internet-based module, PROSPECT
2. Initiation of hormone therapy <4 weeks prior to enrollment in the study
3. Initiation of sleep aids, including over-the-counter or prescription medications taken for insomnia (melatonin, benzodiazepines, antihistamines, etc.) for < 4 weeks prior to enrollment in the study
4. Use of medication for treatment of another sleep disorder, such as restless leg syndrome or narcolepsy
5. History of medial or arthritic disease that could confound or interfere with evaluation of activity level, including but not limited to inflammatory arthritis (Rheumatoid Arthritis, Systemic Lupus Spondyloarthropathy, Psoriatic Arthritis, Polymyalgia Rheumatica), Parkinson's disease and cancer involving the bone
6. Second or third shift workers or others with non-traditional sleep schedules
7. Serious or unstable medical condition that could likely lead to hospitalization during the course of the study or compromise study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | 6 weeks
  Insomnia will be measured through the use of a validated survey called the Insomnia Severity Index

SECONDARY OUTCOMES:
Change in Sleep Disturbance as measured by Actigraphy | 6 weeks
  Sleep disturbance will be measured through the use of actigraphy watches to be worn for 7 days at baseline and 7 days after 6 weeks of the intervention

OTHER OUTCOMES:
Change in use of sleep aids | 6 weeks
  A review of the patient's medication list will be conducted at baseline and 6 weeks to determine change in use of sleep aids for chronic insomnia during study participation
Change in Quality of Life | 6 weeks
  Quality of life will be measured through the use of a validated survey called Functional Assessment of Cancer Therapy-Endocrine Symptoms
Change in Fear of Cancer Recurrence | 6 weeks
  Fear of recurrence will be measured through the use of a validated survey called Assessment of Cancer Survivors

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Hayes, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- Unvisterity of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: For more information about clinical trials at the University of Michigan, including this study — http://www.mcancer.org/about/cancer-answerline